CLINICAL TRIAL: NCT00561730
Title: Pantoprazole 20 mg/40 mg for the Treatment of Gastroesophageal Reflux Disease (GERD)
Brief Title: Efficacy of Pantoprazole in Patients Older Than 12 Years Who Have Symptoms of Non-Erosive Reflux Disease (NERD) or Erosive Gastroesophageal Reflux Disease (eGERD)
Acronym: PANTHER
Status: Completed | Type: Observational
Sponsor: Nycomed (Industry)
Responsible Party: Medical Director, Nycomed Deutschland GmbH
Other Study IDs: PAN 20/40 Panther 07/10
Record Dates: First submitted 2007-11-12; First posted 2007-11-21 (Estimated); Results first posted 2010-09-16 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: PPI (Proton Pump Inhibitor) therapy; Pantoprazole; eGERD (Erosive Gastroesophageal Reflux Disease); NERD (Non-Erosive Reflux Disease)
MeSH Terms: conditions — Gastroesophageal Reflux; Non-Erosive Reflux Disease | interventions — Pantoprazole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pantoprazole: All patients enrolled
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole — Observational, non-interventional study (NIS). The physician decided about dosage according to individual needs (20 or 40 mg pantoprazole, once daily).

SUMMARY:
The aim of the study was to evaluate the effect of 7 days treatment with Pantoprazole 40 mg and 20 mg on symptoms in patients with NERD (non-erosive reflux disease) or eGERD (erosive gastroesophageal reflux disease) in clinical practice. During the study, the patients had to complete a short version of a patient-orientated, self-assessed reflux questionnaire (ReQuest™ in Practice).

ELIGIBILITY:
Main inclusion criteria:

* Outpatients with erosive gastro-esophageal reflux disease (eGERD according to Los Angeles classification grade A-D) or non-erosive reflux disease (NERD)

Main exclusion criteria:

* Criteria as defined in the Summary of Product Characteristics (Chapter 4.3)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatients
Sampling Method: Non-Probability Sample
Enrollment: 1995 (Actual)
Dates: Start 2007-10; Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Thomas D. Bethke, MD, MBA, Study Director — Nycomed Deutschland GmbH, 78467 Konstanz, Germany
Locations (216):
- Germany (216):
  - Nycomed Deutschland GmbH, Aachen
  - Nycomed Deutschland GmbH, Ahrensburg
  - Nycomed Deutschland GmbH, Alfeld
  - Nycomed Deutschland GmbH, Altenburg
  - Nycomed Deutschland GmbH, Altenholz
  - Nycomed Deutschland GmbH, Ansbach
  - Nycomed Deutschland GmbH, Augsburg
  - Nycomed Deutschland GmbH, Bad Bederkesa
  - Nycomed Deutschland GmbH, Bad Bevensen
  - Nycomed Deutschland GmbH, Bad Essen
  - Nycomed Deutschland GmbH, Bad Neustadt an der Saale
  - Nycomed Deutschland GmbH, Bad Säckingen
  - Nycomed Deutschland GmbH, Bad Staffelstein
  - Nycomed Deutschland GmbH, Baden-Baden
  - Nycomed Deutschland GmbH, Beckum
  - Nycomed Deutschland GmbH, Bergisch Gladbach
  - Nycomed Deutschland GmbH, Bergkamen
  - Nycomed Deutschland GmbH, Berlin
  - Nycomed Deutschland GmbH, Bietigheim-Bissingen
  - Nycomed Deutschland GmbH, Bitterfeld-Wolfen
  - Nycomed Deutschland GmbH, Bodenwerder
  - Nycomed Deutschland GmbH, Bonn
  - Nycomed Deutschland GmbH, Brakel
  - Nycomed Deutschland GmbH, Brandenburg
  - Nycomed Deutschland GmbH, Braunschweig
  - Nycomed Deutschland GmbH, Bredstedt
  - Nycomed Deutschland GmbH, Bremen
  - Nycomed Deutschland GmbH, Bremerhaven
  - Nycomed Deutschland GmbH, Buedelsdorf
  - Nycomed Deutschland GmbH, Butzbach
  - Nycomed Deutschland GmbH, Calw
  - Nycomed Deutschland GmbH, Castrop-Rauxel
  - Nycomed Deutschland GmbH, Chemnitz
  - Nycomed Deutschland GmbH, Clausthal-Zellerfeld
  - Nycomed Deutschland GmbH, Cloppenburg
  - Nycomed Deutschland GmbH, Coburg
  - Nycomed Deutschland GmbH, Cologne
  - Nycomed Deutschland GmbH, Cottbus
  - Nycomed Deutschland GmbH, Cölbe
  - Nycomed Deutschland GmbH, Crailsheim
  - Nycomed Deutschland GmbH, Darmstadt
  - Nycomed Deutschland GmbH, Dessau
  - Nycomed Deutschland GmbH, Dinkelsbühl
  - Nycomed Deutschland GmbH, Dinslaken
  - Nycomed Deutschland GmbH, Dortmund
  - Nycomed Deutschland GmbH, Dresden
  - Nycomed Deutschland GmbH, Eisenach
  - Nycomed Deutschland GmbH, Eisenhüttenstadt
  - Nycomed Deutschland GmbH, Ellefeld
  - Nycomed Deutschland GmbH, Engelskirchen
  - Nycomed Deutschland GmbH, Erfurt
  - Nycomed Deutschland GmbH, Eschweiler
  - Nycomed Deutschland GmbH, Essen
  - Nycomed Deutschland GmbH, Flensburg
  - Nycomed Deutschland GmbH, Frankenberg
  - Nycomed Deutschland GmbH, Frankenthal
  - Nycomed Deutschland GmbH, Frankfurt
  - Nycomed Deutschland GmbH, Freiburg im Breisgau
  - Nycomed Deutschland GmbH, Freising
  - Nycomed Deutschland GmbH, Freudenstadt
  - Nycomed Deutschland GmbH, Fulda
  - Nycomed Deutschland GmbH, Fürth
  - Nycomed Deutschland GmbH, Gaggenau
  - Nycomed Deutschland GmbH, Garbsen
  - Nycomed Deutschland GmbH, Gelsenkirchen
  - Nycomed Deutschland GmbH, Genthin
  - Nycomed Deutschland GmbH, Gera
  - Nycomed Deutschland GmbH, Goch
  - Nycomed Deutschland GmbH, Göppingen
  - Nycomed Deutschland GmbH, Göttingen
  - Nycomed Deutschland GmbH, Greiz
  - Nycomed Deutschland GmbH, Gresse
  - Nycomed Deutschland GmbH, Grevenbroich
  - Nycomed Deutschland GmbH, Grevesmühlen
  - Nycomed Deutschland GmbH, Güstrow
  - Nycomed Deutschland GmbH, Halberstadt
  - Nycomed Deutschland GmbH, Halle
  - Nycomed Deutschland GmbH, Hamburg
  - Nycomed Deutschland GmbH, Hanover
  - Nycomed Deutschland GmbH, Hardheim
  - Nycomed Deutschland GmbH, Harra
  - Nycomed Deutschland GmbH, Haßloch
  - Nycomed Deutschland GmbH, Hechingen
  - Nycomed Deutschland GmbH, Heide
  - Nycomed Deutschland GmbH, Henstedt-Ulzburg
  - Nycomed Deutschland GmbH, Herford
  - Nycomed Deutschland GmbH, Herne
  - Nycomed Deutschland GmbH, Herrieden
  - Nycomed Deutschland GmbH, Hildesheim
  - Nycomed Deutschland GmbH, Hof
  - Nycomed Deutschland GmbH, Hofbieber
  - Nycomed Deutschland GmbH, Johanngeorgenstadt
  - Nycomed Deutschland GmbH, Karlstadt am Main
  - Nycomed Deutschland GmbH, Kassel
  - Nycomed Deutschland GmbH, Kelkheim
  - Nycomed Deutschland GmbH, Kiel
  - Nycomed Deutschland GmbH, Koblenz
  - Nycomed Deutschland GmbH, Kornwestheim
  - Nycomed Deutschland GmbH, Köthen
  - Nycomed Deutschland GmbH, Kronach
  - Nycomed Deutschland GmbH, Künzing
  - Nycomed Deutschland GmbH, Landstuhl
  - Nycomed Deutschland GmbH, Lebach
  - Nycomed Deutschland GmbH, Leinfelden-Echterdingen
  - Nycomed Deutschland GmbH, Leipzig
  - Nycomed Deutschland GmbH, Leisnig
  - Nycomed Deutschland GmbH, Leverkusen
  - Nycomed Deutschland GmbH, Lichtenfels
  - Nycomed Deutschland GmbH, Lingen
  - Nycomed Deutschland GmbH, Ludwigsburg
  - Nycomed Deutschland GmbH, Ludwigsfelde
  - Nycomed Deutschland GmbH, Ludwigshafen
  - Nycomed Deutschland GmbH, Ludwigslust
  - Nycomed Deutschland GmbH, Lübeck
  - Nycomed Deutschland GmbH, Lüdenscheid
  - Nycomed Deutschland GmbH, Lüneburg
  - Nycomed Deutschland GmbH, Lützen
  - Nycomed Deutschland GmbH, Magdeburg
  - Nycomed Deutschland GmbH, Mainz
  - Nycomed Deutschland GmbH, Mannheim
  - Nycomed Deutschland GmbH, Marburg
  - Nycomed Deutschland GmbH, Marienberg
  - Nycomed Deutschland GmbH, Marl
  - Nycomed Deutschland GmbH, Mayen
  - Nycomed Deutschland GmbH, Merseburg
  - Nycomed Deutschland GmbH, Merzig
  - Nycomed Deutschland GmbH, Minden
  - Nycomed Deutschland GmbH, Möckmühl
  - Nycomed Deutschland GmbH, Mönchengladbach
  - Nycomed Deutschland GmbH, München
  - Nycomed Deutschland GmbH, Münzenberg
  - Nycomed Deutschland GmbH, Neckargemünd
  - Nycomed Deutschland GmbH, Neu Wulmstorf
  - Nycomed Deutschland GmbH, Neu-Isenburg
  - Nycomed Deutschland GmbH, Neubiberg
  - Nycomed Deutschland GmbH, Neukirchen
  - Nycomed Deutschland GmbH, Neustadt
  - Nycomed Deutschland GmbH, Neuwied
  - Nycomed Deutschland GmbH, Nieder-Olm
  - Nycomed Deutschland GmbH, Nienburg
  - Nycomed Deutschland GmbH, Nordhorn
  - Nycomed Deutschland GmbH, Nuremberg
  - Nycomed Deutschland GmbH, Oberhausen
  - Nycomed Deutschland GmbH, Oberndorf
  - Nycomed Deutschland GmbH, Ochsenfurt
  - Nycomed Deutschland GmbH, Oelsnitz
  - Nycomed Deutschland GmbH, Oschatz
  - Nycomed Deutschland GmbH, Oschersleben
  - Nycomed Deutschland GmbH, Osnabrück
  - Nycomed Deutschland GmbH, Paderborn
  - Nycomed Deutschland GmbH, Papenburg
  - Nycomed Deutschland GmbH, Peine
  - Nycomed Deutschland GmbH, Penig
  - Nycomed Deutschland GmbH, Pfullingen
  - Nycomed Deutschland GmbH, Pirna
  - Nycomed Deutschland GmbH, Plauen
  - Nycomed Deutschland GmbH, Potsdam
  - Nycomed Deutschland GmbH, Recklinghausen
  - Nycomed Deutschland GmbH, Regensburg
  - Nycomed Deutschland GmbH, Reichenbach
  - Nycomed Deutschland GmbH, Remscheid
  - Nycomed Deutschland GmbH, Rendsburg
  - Nycomed Deutschland GmbH, Reutlingen
  - Nycomed Deutschland GmbH, Riesa
  - Nycomed Deutschland GmbH, Roetgen
  - Nycomed Deutschland GmbH, Rostock
  - Nycomed Deutschland GmbH, Rottach-Egern
  - Nycomed Deutschland GmbH, Rottweil
  - Nycomed Deutschland GmbH, Saarbrücken
  - Nycomed Deutschland GmbH, Saarlouis
  - Nycomed Deutschland GmbH, Saint Blasien
  - Nycomed Deutschland GmbH, Salzgitter
  - Nycomed Deutschland GmbH, Salzmünde
  - Nycomed Deutschland GmbH, Sangerhausen
  - Nycomed Deutschland GmbH, Sarstedt
  - Nycomed Deutschland GmbH, Schiffweiler
  - Nycomed Deutschland GmbH, Schmalkalden
  - Nycomed Deutschland GmbH, Schönwalde-Glien
  - Nycomed Deutschland GmbH, Schwäbisch Hall
  - Nycomed Deutschland GmbH, Schwedt
  - Nycomed Deutschland GmbH, Schwerin
  - Nycomed Deutschland GmbH, Siegen
  - Nycomed Deutschland GmbH, Sinsheim
  - Nycomed Deutschland GmbH, Spaichingen
  - Nycomed Deutschland GmbH, Steinfurt
  - Nycomed Deutschland GmbH, Steißlingen
  - Nycomed Deutschland GmbH, Stockach
  - Nycomed Deutschland GmbH, Strausberg
  - Nycomed Deutschland GmbH, Stuhr
  - Nycomed Deutschland GmbH, Sundern
  - Nycomed Deutschland GmbH, Teuchern
  - Nycomed Deutschland GmbH, Tönisvorst
  - Nycomed Deutschland GmbH, Travemünde
  - Nycomed Deutschland GmbH, Trier
  - Nycomed Deutschland GmbH, Trittau
  - Nycomed Deutschland GmbH, Varel
  - Nycomed Deutschland GmbH, Waghäusel
  - Nycomed Deutschland GmbH, Wangen
  - Nycomed Deutschland GmbH, Wanzleben
  - Nycomed Deutschland GmbH, Wäschenbeuren
  - Nycomed Deutschland GmbH, Weißwasser
  - Nycomed Deutschland GmbH, Westerkappeln
  - Nycomed Deutschland GmbH, Weyhe
  - Nycomed Deutschland GmbH, Wiesbaden
  - Nycomed Deutschland GmbH, Wiesloch
  - Nycomed Deutschland GmbH, Willich
  - Nycomed Deutschland GmbH, Winsen
  - Nycomed Deutschland GmbH, Wismar
  - Nycomed Deutschland GmbH, Wittenberg
  - Nycomed Deutschland GmbH, Wittstock
  - Nycomed Deutschland GmbH, Wolfsburg
  - Nycomed Deutschland GmbH, Worms
  - Nycomed Deutschland GmbH, Würzburg
  - Nycomed Deutschland GmbH, Zerbst
  - Nycomed Deutschland GmbH, Zweibrücken
  - Nycomed Deutschland GmbH, Zwickau

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pantoprazole
Started | 1995
Completed | 1986
Not Completed | 9
Not completed — Adverse Event | 2
Not completed — Handling of the drug | 1
Not completed — Lost to Follow-up | 5
Not completed — Not specified reasons | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pantoprazole
Number analyzed (Participants) | 1995
Age Continuous [Mean (Standard Deviation); unit: Years] — The measured value is related to the number of 1977 subjects (= valid cases). This number differs from the overall number of baseline participants due to missing data for 18 subjects.
  Years | 54.1 (15.0)
Sex/Gender, Customized [Number; unit: Percentage of participants]
  Female | 46.3
  Male | 53.4
  Missing data | 0.3
Nicotine use [Number; unit: Percentage of participants]
  Smoker | 32.5
  Non-smoker | 66.8
  Missing data | 0.7
Alcohol use [Number; unit: Percentage of participants]
  Daily | 17.3
  Not daily | 82.2
  Missing data | 0.5
Drug abuse [Number; unit: Percentage of participants]
  Drug abuse | 1.0
  No drug abuse | 98.0
  Missing data | 1.0
Diagnosis: reflux disease [Number; unit: Percentage of participants]
  Non-Erosive Reflux Disease (NERD) | 35.1
  Erosive Gastroesophageal Reflux Disease (eGERD) | 64.1
  Missing data | 0.9

OUTCOME MEASURES:

1. Primary Outcome: Patient's Assessment of General Well-being During the Last 24 Hours (Diaries; ReQuest™ in Practice)
Description: Assessment on a scale: Severity from 0=Excellent to 10=Extremely bad
Time Frame: 7 days
Population: All patients included and treated, intention to treat, missing values not imputed ('as observed').
  Number of valid cases:
  * Day 0 = 1769
  * Day 1 = 1760
  * Day 2 = 1761
  * Day 3 = 1751
  * Day 4 = 1749
  * Day 5 = 1742
  * Day 6 = 1747
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Pantoprazole: All patients with valid value at least at day 0
Arm/Group | Pantoprazole
Number analyzed (Participants) | 1769
Units on a scale
  Day 0 | 5.31 (2.27)
  Day 1 | 4.60 (2.26)
  Day 2 | 3.67 (2.08)
  Day 3 | 2.95 (1.94)
  Day 4 | 2.51 (1.82)
  Day 5 | 2.14 (1.70)
  Day 6 | 1.91 (1.63)

2. Primary Outcome: Patient's Assessment of Acid Complaints During the Last 24 Hours (Diaries; ReQuest™ in Practice)
Description: Assessment on a scale: Severity from 0=None to 10=Extremely strong
Time Frame: 7 days
Population: All patients included and treated, intention to treat, missing values not imputed ('as observed').
  Number of valid cases:
  * Day 0 = 1767
  * Day 1 = 1758
  * Day 2 = 1757
  * Day 3 = 1744
  * Day 4 = 1743
  * Day 5 = 1739
  * Day 6 = 1739
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 1767
Units on a scale
  Day 0 | 6.14 (2.46)
  Day 1 | 4.62 (2.45)
  Day 2 | 3.34 (2.16)
  Day 3 | 2.43 (1.83)
  Day 4 | 1.94 (1.59)
  Day 5 | 1.57 (1.36)
  Day 6 | 1.33 (1.22)

3. Primary Outcome: Patient's Assessment of Upper Abdominal/Stomach Complaints During the Last 24 Hours (Diaries; ReQuest™ in Practice)
Description: Assessment on a scale: Severity from 0=None to 10=Extremely strong
Time Frame: 7 days
Population: All patients included and treated, intention to treat, missing values not imputed ('as observed').
  Number of valid cases:
  * Day 0 = 1760
  * Day 1 = 1750
  * Day 2 = 1746
  * Day 3 = 1735
  * Day 4 = 1735
  * Day 5 = 1730
  * Day 6 = 1734
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 1760
Units on a scale
  Day 0 | 4.73 (2.57)
  Day 1 | 3.66 (2.33)
  Day 2 | 2.71 (2.02)
  Day 3 | 2.11 (1.73)
  Day 4 | 1.75 (1.51)
  Day 5 | 1.49 (1.32)
  Day 6 | 1.31 (1.25)

4. Primary Outcome: Patient's Assessment of Lower Abdominal/Digestive Complaints During the Last 24 Hours (Diaries; ReQuest™ in Practice)
Description: Assessment on a scale: Severity from 0=None to 10=Extremely strong
Time Frame: 7 days
Population: All patients included and treated, intention to treat, missing values not imputed ('as observed').
  Number of valid cases:
  * Day 0 = 1754
  * Day 1 = 1742
  * Day 2 = 1739
  * Day 3 = 1733
  * Day 4 = 1730
  * Day 5 = 1726
  * Day 6 = 1729
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 1754
Units on a scale
  Day 0 | 2.48 (2.21)
  Day 1 | 2.12 (1.96)
  Day 2 | 1.76 (1.72)
  Day 3 | 1.52 (1.48)
  Day 4 | 1.40 (1.42)
  Day 5 | 1.27 (1.31)
  Day 6 | 1.20 (1.26)

5. Primary Outcome: Patient's Assessment of Nausea During the Last 24 Hours (Diaries; ReQuest™ in Practice)
Description: Assessment on a scale: Severity from 0=None to 10=Extremely strong
Time Frame: 7 days
Population: All patients included and treated, intention to treat, missing values not imputed ('as observed').
  Number of valid cases:
  * Day 0 = 1755
  * Day 1 = 1744
  * Day 2 = 1742
  * Day 3 = 1728
  * Day 4 = 1727
  * Day 5 = 1724
  * Day 6 = 1726
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 1755
Units on a scale
  Day 0 | 3.00 (2.54)
  Day 1 | 2.38 (2.14)
  Day 2 | 1.84 (1.77)
  Day 3 | 1.51 (1.45)
  Day 4 | 1.30 (1.29)
  Day 5 | 1.13 (1.13)
  Day 6 | 1.02 (0.96)

6. Primary Outcome: Patient's Assessment of Sleep Disturbances During the Last 24 Hours (Diaries; ReQuest™ in Practice)
Description: Assessment on a scale: Severity from 0=None to 10=Extremely strong
Time Frame: 7 days
Population: All patients included and treated, intention to treat, missing values not imputed ('as observed').
  Number of valid cases:
  * Day 0 = 1755
  * Day 1 = 1740
  * Day 2 = 1740
  * Day 3 = 1733
  * Day 4 = 1732
  * Day 5 = 1725
  * Day 6 = 1727
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 1755
Units on a scale
  Day 0 | 3.15 (2.68)
  Day 1 | 2.62 (2.36)
  Day 2 | 2.15 (2.05)
  Day 3 | 1.85 (1.83)
  Day 4 | 1.62 (1.64)
  Day 5 | 1.49 (1.54)
  Day 6 | 1.38 (1.42)

7. Secondary Outcome: Physician's Assessment of Heartburn
Description: Assessment on a scale: 1=none, 2=mild, 3=moderate, 4=severe
Time Frame: 7 days
Population: Patients included and treated with valid data at first and last visit (without imputation of missing values), intention to treat
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Pantoprazole: All patients with valid values at first and last visit
Arm/Group | Pantoprazole
Number analyzed (Participants) | 1960
Units on a scale
  Start of therapy | 3.08 (0.76)
  End of study | 1.35 (0.57)

8. Secondary Outcome: Physician's Assessment of Acid Eructation
Description: Assessment on a scale: 1=none, 2=mild, 3=moderate, 4=severe
Time Frame: 7 days
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 1950
Units on a scale
  Start of therapy | 2.74 (0.85)
  End of study | 1.25 (0.52)

9. Secondary Outcome: Physician's Assessment of Painful Swallowing
Description: Assessment on a scale: 1=none, 2=mild, 3=moderate, 4=severe
Time Frame: 7 days
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 1945
Units on a scale
  Start of therapy | 1.72 (0.84)
  End of study | 1.07 (0.30)

10. Secondary Outcome: Assessment of the Efficacy of Pantoprazole 20 mg/40 mg at Final Visit
Description: Assessment on a scale: 1=excellent, 2=good, 3=satisfactory, 4=not satisfactory
Time Frame: 7 days
Population: Patients included and treated with at least one application of pantoprazole (without imputation of missing values), intention to treat
Measure: Number; unit: Percentage of participants
Groups:
- Pantoprazole: Patients included and treated with at least one application of pantoprazole
Arm/Group | Pantoprazole
Number analyzed (Participants) | 1995
Percentage of participants
  Excellent | 67.4
  Good | 25.0
  Satisfactory | 3.0
  Not satisfactory | 0.7
  Missing data | 3.9

11. Secondary Outcome: Assessment of the Tolerability of Pantoprazole 20 mg/40 mg at Final Visit
Description: Assessment on a scale: 1=excellent, 2=good, 3=satisfactory, 4=not satisfactory
Time Frame: 7 days
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Pantoprazole
Number analyzed (Participants) | 1995
Percentage of participants
  Excellent | 81.1
  Good | 14.0
  Satisfactory | 1.0
  Not satisfactory | 0.1
  Missing data | 3.9

ADVERSE EVENTS:
Time Frame: First until last visit (planned 7 days)
Arm/Group | Pantoprazole
Serious Adverse Events (participants affected / at risk) | 1/1995
Other Adverse Events (participants affected / at risk) | 10/1995
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pantoprazole (N=1995)
Nervousness (Psychiatric disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.01% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pantoprazole (N=1995)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Flatulence (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 2 (2)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No